CLINICAL TRIAL: NCT04950088
Title: Reduction of Perioperative Anxiety Using a Hand-held Video Game Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00057182
Record Dates: First submitted 2021-06-22; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Separation Anxiety; Anxiety; Anxiety, Separation; Anxiety Generalized
Keywords: anxiety; separation fear
MeSH Terms: conditions — Anxiety, Separation; Anxiety Disorders; Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: Patients will be assigned into a "Video Game group" or a "No Video Game group." All patients on any particular day will be assigned into the same group. This is done to prevent one patient from feeling disappointed after seeing another patient with a video game, and then learning they may not have one. Group assignment will alternate each day.
Who Masked: Participant, Care Provider
Masking Description: participants didn't know if it was 'game day' or 'no game day' but were consented to fill out surveys regardless of the status of game day. Care providers provided games on game day or didn't provide games on 'no game day' but didn't have foreknowledge of which participants had consented to the study until they reached the peri-operative suite.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game (Active Comparator): Patients will be assigned into a "Video Game group" or a "No Video Game group." All patients on any particular day will be assigned into the same group. This is done to prevent one patient from feeling disappointed after seeing another patient with a video game, and then learning they may not have one. Group assignment will alternate each day.
  Interventions: Other: Hand-held video game device
- no game (Active Comparator): Patients will be assigned into a "Video Game group" or a "No Video Game group." All patients on any particular day will be assigned into the same group. This is done to prevent one patient from feeling disappointed after seeing another patient with a video game, and then learning they may not have one. Group assignment will alternate each day.
  Interventions: Other: Hand-held video game device

INTERVENTIONS:
Other: Hand-held video game device

SUMMARY:
Distraction techniques, such as use of a virtual reality device, have been used to augment or replace pharmacological practices for relief of anxiety in pediatric patients prior to surgical procedures. This relief can not only benefit medical staff, as procedures may be easier to perform and require less time, but also have a calming effect on the the parent during the procedure if they feel that their child is being better cared for. In addition, decreased anxiety prior to surgical procedures have been shown to reduce maladaptive behaviors post-operatively. This prospective study plans to evaluate the anxiety level of parents and pediatric patients in an outpatient surgery center pre-, during and post-operatively with and without the use of a virtual reality distraction device. The goal is to determine the existence of correlations between distraction techniques (in this case, the use of handheld video games) pediatric patient anxiety, parental anxiety, and parental satisfaction with the experience surrounding the procedure.

DETAILED DESCRIPTION:
General Data will be collected for patients being treated at Patewood Outpatient Surgery Center following legal guardian consent. Patients receiving surgical treatment involving the use of an anesthesia mask, age 4 to 10, will be included in the study. Exclusion criteria will include ear tube cases, patients physically incapable to play a video game, patients of non-English speaking caregivers, and patients without legal guardian present day of surgery. IV Ear tube cases are too short a procedure for data collection and at least one caretaker must be capable of taking both an oral and written survey.

For the purposes of this study, a "caregiver" will be defined as an adult that spends a significant amount of time with the patient, and meets the following criteria.

The primary caregiver is the adult that is responsible for the minor patients' care. The caregiver may reside with the patient full-time or part-time but have the information necessary to assess the child's behavior before and after the outpatient procedure.

Data collected for each patient will include demographics, random placement in Video Game/No Video game group, surgical procedure, information normally recorded by surgeon or anesthesiologist including duration of surgery and duration under anesthesia, caregiver reported changes in patient behavior following surgery, and scores of the anxiety being felt by caregivers and patients. Anxiety scores will be determined using shortened versions of validated anxiety scoring assessments. Behavioral changes will be recorded using a shortened version of the Post Hospital Behavior Questionnaire (PHBQ). Assessments have been shortened to increase study participation, and eliminate any impact the study may have had on day-to-day operations at Patewood Outpatient Surgery Center.

Caregivers will also be asked to fill out a hospital created survey related to how satisfied they are with the care of the patient. It will be referred to as the Preoperative Hospital Satisfaction Survey (PHSS). This survey will be administered while the surgical procedure is in progress, when the caregivers are sitting in the waiting room. The survey is to be a reflection of how caregivers perceive preoperative separation care given to patients, so will not be influenced by surgical outcome.

Consent Legal guardians of patients are contacted over the phone by Patewood Outpatient Surgery Center registration per standard preoperative care procedure. Before concluding the normal preoperative interview, a script will be read that introduces the guardian to the study and its goals. The guardian will then be asked if they are interested in learning more about the study. Those who answer "no" will be removed from a list of potential participants. Those who answer "yes" or "maybe" will be given more information about study participation after arriving at the outpatient surgery center on the day of their scheduled appointment. A more thorough explanation of the study will be given and any questions answered. If a guardian is interested in participating, they will be provided a consent form to fill out.

Group assignment Patients will be assigned into a "Video Game group" or a "No Video Game group." All patients on any particular day will be assigned into the same group. This is done to prevent one patient from feeling disappointed after seeing another patient with a video game, and then learning they may not have one. Group assignment will alternate each day.

Assessment and Survey Descriptions

Modified Yale Preoperative Scale (mYPAS)- Observational survey used to quickly score the anxiety level of children during preoperative holding and induction of anesthesia. It has frequent use and validation as an accurate tool for determining the anxiety level of pediatric surgical patients. Each section has 4 to 6 numbers listed, each corresponding with different patient description. For each section, the number by the most accurate patient description is circled. (Jenkins)(Kain)

State Trait Anxiety Inventory (STAI)- Self-taken survey for adults. Gives 2 different scores. One score is an indicator of susceptibility to stressful situations, the other score is the level of anxiety felt while taking the survey. It has frequent use and validation as a tool for determining anxiety levels of adults. (Spielberger)

Post Hospital Behavior Questionnaire (PHBQ)- Survey taken by primary caregiver of a patient after leaving the hospital. The survey is designed to identify maladaptive behaviors a patient has developed following a time at a hospital. Questions must be answered "much less than before", "less than before", "same as before", "more than before", or "much more than before". This survey is sensitive only to the change in frequency of behaviors, not their presence or absence. Therefore, undesirable behavior existing prior to a hospital stay should have no influence on the PHBQ score.

All surveys used in this study were truncated. Any modification was evaluated and approved by the staff psychologist (PhD.) familiar with using surveys to research anxiety and stress of patients and their families. Any questions that were included or excluded from the surveys was done so under expert direction.

Perioperative Holding After completing standard preoperative procedure, a nurse will complete a short observational survey (mYPAS [modified Yale Preoperative Scale] or mYPAS-SF) to score the patients current anxiety level. Just prior to separation from the caregiver, the patient will be given (or not given) a Video Game by the nurse. During separation, another mYPAS will be scored.

Operating Room Another mYPAS will be scored during the induction of anesthesia. If the patient has a video game, the patient is allowed to play as long as he/she wants. Often times, this is up until the procedure begins.

Caregivers During Procedure One or two primary caregivers will be asked to fill out a shortened STAI (State Trait Anxiety Inventory) and PHSS.

Follow-up Phone Calls The day following surgery, standard postoperative care procedure will be followed. This includes a phone call to the caregiver of a patient. Before concluding the phone call, the instructions at the top of the shortened PHBQ will be read to the caregivers participating in the survey. Then each question will be read and answered. One week and 2 weeks following surgery, the caregiver will be called and the shortened PHBQ will be administered.

Statistics The existence of correlations between maladaptive behavior, patient anxiety, caregiver susceptibility to anxiety, caregiver experience of anxiety, caregiver satisfaction, video game use, and any other collected data will be determined. All information from this study will be used to describe our cohort only. All data will be expressed in summary and is meant to contribute to the generalizable knowledge of the field.

ELIGIBILITY:
Inclusion Criteria:

* outpatient pediatric surgery patients between July 2016 and October 2016.
* Children, (ages 3-10 years) undergoing low-risk outpatient surgical procedures, including, but not limited to, tonsillectomies, adenoidectomies, etc., for which a masked induction was planned
* guardians of the children had to be present and consent.

Exclusion Criteria:

* patients undergoing ear tube placement/removal (due to the short duration of the procedure)
* patients requiring premedication
* patients with physical or mental disabilities rendering it difficult to use the distraction device
* non-English speaking caregivers (due to the language barriers during the post-operative phone calls).
* patients without guardians providing consent

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in pediatric anxiety score | at three timepoints in the peri-operative suite prior to induction for surgery
  The modified Yale Preoperative Anxiety Scale16 (mYPAS): evaluated changes in pediatric anxiety with higher anxiety=higher score. mYPAS completed by nurses during initial preoperative evaluation, upon patient separation from parent and at mask induction. All three surveys were identical.
  A. Activity scored 1-4; B. Vocalizations scored 1-6; C. Emotional expressivity scored 1-4; D. State of apparent arousal scored 1-4
Change in parent anxiety score | Immediately following separation from the child; change in anxiety from baseline
  The Strait-Trait Anxiety Inventory (STAI)17 assessed self-reported parental anxiety (below). The STAI was completed by the parent immediately after separation in the waiting room. STAI consists of two parts: A= perceived anxiety during the child's perioperative period; B= the parent's general state of anxiety. Differences between these two metrics were used to indicate parental satisfaction with their experience.
  The A questions were evaluated with the following scale (1-4) utilizing the descriptors
  'Not at all' 'Somewhat' 'Moderately So' 'Very Much So' in response to 7 statements.
  The B section regarding generalized anxiety was measured as follows (1-4) utilizing the descriptors
  'Not at all' 'Somewhat' 'Moderately So' 'Very Much So' in response to 7 statements different from the A section.
  The final question is as follows (Y/N):
  8. The experience of separation from my child for this procedure was better than expected. Y N
Overall Parental Satisfaction with the pre-operative process, particularly regarding parent/child separation | Immediately following separation from the child
  To evaluate overall satisfaction of parents with the pre-operative process specifically, a final question was added to the STAI which inquired if the parent/guardian thought that the experience of separation was better or worse than was expected. This question was scored independently.
Change in post-operative behavior as assessed by the parent | 24-48 hours, 7 days and 14 days post procedure
  The PHBQ queried change in perceived patient's behavior before and after the procedure with an inquiry regarding new-onset negative behaviors manifesting post-surgery. Three attempts were made to gather survey information for each time-point; if a parent could not be reached, data collection for that patient was truncated. Each of the three follow-up calls were completed utilizing the same protocol. The protocol consisted of 10 questions regarding the child's behavior with parent answers utilizing the following scale:
  much less less same more much more
  The final question was a rank from 1-10 with 10 being the worst (highest) score:
  11. On a scale from 1 to 10, 1 being no pain and 10 being more pain, how would you rate your child's current pain level?
  1 2 3 4 5 6 7 8 9 10